CLINICAL TRIAL: NCT04574271
Title: Multidimensional Intervention Directed to Pre-frail Patients Older Than 70 Years from Primary Care in a Basic Semi-urban Health Area
Brief Title: Multidimensional Intervention in Pre-frail Patients Older Than 70 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endocrinology and Clinical Nutrition Research Center, Spain (Other)
Responsible Party: Principal Investigator, Daniel de Luis Roman, Professor, MD, PhD, Endocrinology and Clinical Nutrition Research Center, Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI 19-1425
Record Dates: First submitted 2020-09-27; First posted 2020-10-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Frail Elderly Syndrome; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: * Intervention Group: Intensitve nutritional advice and exercise prescription adapted to physical performance.
  * Control Group: Usual nutritional advice and exercise prescription.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive dietary advice and exercise prescription (Experimental): Personalized dietary advice and exercise prescription according to nutritional status.
  Interventions: Behavioral: Intensive dietary advice and exercise prescription
- Usual dietary advice and exercise prescription (Active Comparator): Generalized dietary advice and exercise prescription in elder subjects.
  Interventions: Behavioral: Usual dietary advice and exercise prescription

INTERVENTIONS:
Behavioral: Intensive dietary advice and exercise prescription — Personalized dietary advice and exercise prescription according to nutritional status.
  Other Names: Personalized dietary advice and exercise prescription
  Arms: Intensive dietary advice and exercise prescription
Behavioral: Usual dietary advice and exercise prescription — Generalized dietary advice and excercise prescription in elder patients.
  Arms: Usual dietary advice and exercise prescription

SUMMARY:
Aging represents a huge advance in society and a health and social challenge. Spain has one of the highest life expectancies in the world, but other countries with the same demographic characteristics are ahead of us in quality adjusted life years. Primary care setting has the main drivers of healthy aging, acting on the early stages of pre-frailty and frailty.

Therefore, it is proposed a multicomponent intervention (nutritional and prescription of physical exercise) in patients older than 70 years of the Medina del Campo Health Center, with pre-frailty criteria, in order to measure the changes that this intervention produces in their mild dysfunction and whether it is capable of reversing it or delaying the progression to a state of frailty.

DETAILED DESCRIPTION:
Hypothesis: A balanced diet, with a sufficient protein intake for each patient based on the Mediterranean diet, as well as the performance of multicomponent exercise 3 times a week, delays the evolution to stages of dysfunction or disability in the pre-frail population.

Objective:

* The main objective is to evaluate the effect of an intensive nutritional dietary treatment on the function markers in a sample of elderly people in a situation of pre-frailty.
* To Demonstrate the equivalence of the values obtained in terms of functional improvement through adequate exercise and diet in urban populations in a semi-urban population.
* To evaluate the change in analytical markers that indicate pre-frailty in patients under intensive dietary-nutritional treatment.
* To Study the improvement of quality of life in individuals with adequate nutrition and level of physical exercise in those over 70 years of age in pre-frailty stages, increasing the prevalence of healthy aging in our study population.

Methods:

- Design: This is a quasi-experimental study with a control group. Recruitment will be carried out, through random sampling, of patients over 70 years of age from the basic health area of Medina del Campo Urbano, detecting those who meet Fried's pre-frailty criteria, through the FRAIL questionnaire, being positive for pre-frailty fulfilling 1 or 2 criteria. These subjects detected as pre-frail will be randomly included in different multicomponent programs. In a group, two types of interventions will be carried out by the research team from primary care: Dietary advice adjusted to the needs of the patient and their pre-frailty stage, with an adequate nutritional and protein intake, based on the scientific evidence existing to date and in collaboration with the Clinical Hospital of Valladolid, Spain; and a multicomponent physical exercise prescription (elasticity, strength, resistance and balance), of at least 150 minutes per week, according to the WHO recommendations for this age group, adapting it individually, to be performed 3-5 times per week. Both branches of the intervention will be carried out through periodic interviews throughout a year of follow-up.

In the control group, the nutritional advice and prescription of regular physical exercise will be developed by the health team of the primary care center.

During this year, the parameters to be measured of functionality and independence, as well as anthropometric, quality of life and corresponding analytical parameters will be evaluated prior to the beginning of the intervention. Evaluating their variation at 3 months, 6 months and one year in both groups.

* Sample Size: It has been calculated to estimate a proportion similar to that of the population. Based on the prevalence of 50% existing in other study samples in the national territory for pre-frailty, and thus choosing the position of maximum indeterminacy (p = 50), assuming normality, for an α = 0.05 the Measure of the resulting sample calculated was 338 individuals.
* Chronogram:

Selection of patients: june 2019. Phone recruiting of patients: june 2019 Clinical and functional assessment will be carried out in Medina del Campo Health Center and randomization: july 2019-August 2019.

Intervention (First Time): October-december 2019; january-february 2020; july-august 2020; september-october 2020.

Follow up: Evaluation of parameters. July-August 2020; september-october 2020; november-december 2020; january-february 2021.

Statistycal Analysis: March-April 2021 Drafting of results: May-June 2021

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized patients over 70 years of age from the basic health area of Medina del Campo Urbano, who meet pre-frailty criteria (1 or 2 Fried criteria).

Exclusion Criteria:

* Cognitive impairment
* Frailty syndrome
* Moderate-Severe Dependence
* Life Expectancy less than 6 months or patients in palliative care

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 340 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Functional assessment by Fried Criteria | 12 months
  Test of frail syndrome diagnosis in elder patients (Three out five criteria)
Fall Risk by test up and go | 12 months
  Functional tests of frail syndrome diagnosis in elder patients (<10 seconds: low fall risk; 10-20 seconds: fragility (risk of fall); >20 seconds: high risk of fall).
The Lawton Instrumental Activities of Daily Living (IADL) Scale | 12 months
  Functional tests of frail syndrome diagnosis in elder patients (Grade of depedence: <20: Total; 20-35: Severe; 40-55: Moderate; >60: Mild; 100: Independent).
Barthel Test for dependency | 12 months
  Functional tests of frail syndrome diagnosis in elder patients

SECONDARY OUTCOMES:
Mini-Mental Test | 12 months
  Cognitive evaluation (0-14: severe cognitive impairment; 15-19: moderate cognitive impairment; 20-24 mild cognitive impairment; 25-30: soft deficit of cognitive function; 30-35: normal).
Short Form 36 (SF-36) Health survey Questionnaire | 12 months
  Questionnaire to measure quality of life (0-100 --> 0=worst health status - 100=better health status).

CONTACTS AND LOCATIONS:
Overall Officials: Juan J LOPEZ-GOMEZ, MD; PhD, Principal Investigator — Hospital Clínico Universitario de Valladolid; Daniel A De Luis Román, MD; PhD, Study Director — University of Valladolid; Cristina Gutiérrez-Lora, MD, Principal Investigator — Primary Care Center (Medina del Campo (Valladolid, Spain))
Locations (1):
- Cristina Gutiérrez-Lora, Medina del Campo, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No